CLINICAL TRIAL: NCT00159432
Title: Phase II Study of Oxaliplatin, Capecitabine and Bevacizumab as First Line Treatment for Patients With Advanced Colorectal Cancer
Brief Title: Study of Oxaliplatin, Capecitabine and Bevacizumab as First Line Treatment for Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Hoffmann-La Roche (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-04-10
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal; cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Oxaliplatin; Bevacizumab; Capecitabine

ARMS (1):
- Oxaliplatin, followed by Bevacizumab with Capecitabine (Experimental): oxaliplatin 85 mg/m2 q 14 days, followed by bevacizumab 5 mg/kg q 14 days, with capecitabine 750 mg/m2 bid daily
  Interventions: Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: Bevacizumab
  Other Names: Avastin
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
This study is for people with colorectal cancer, who have tumors that cannot be completely removed by surgery. This study is being done to find out how long it takes tumors to grow after patients receive the drugs capecitabine, oxaliplatin and bevacizumab. Capecitabine (also called Xeloda) is a drug that has been approved by the FDA for treatment of advanced colorectal cancer. Capecitabine prevents some colorectal cancer cancer cells from reproducing, and causes some of them to die. Oxaliplatin (also called Eloxatin) has also been approved by the FDA for treatment of advanced colorectal cancer. Oxaliplatin prevents some colorectal cancer cells from reproducing. Bevacizumab is an investigational drug. Bevacizumab is an antibody (a protein that acts against a specific substance) directed against vascular endothelial growth factor (VEGF). VEGF promotes the growth of blood vessels that bring nutrients to cells. Bevacizumab inhibits the growth of colon cancer cells, by blocking the effects of VEGF. The combination of the drugs used in this study is experimental. The purpose of this study is to see how long it takes patients' tumors to grow when they are taking this combination of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or recurrent colorectal tumors with no previous treatment for advanced disease.
* Age greater than or equal to 18 years
* SWOG performance status 0-1.
* At least one measurable lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques.
* Have a negative serum pregnancy test within 7 days prior to initiation of chemotherapy (female patients of childbearing potential).
* Availability of tumor biopsy (paraffin embedded or fresh frozen) at the time of diagnosis and/or prior to study entry is required.
* Patients must agree to have a 20 cc blood sample drawn in addition to routine labs with each cycle of chemotherapy.

Exclusion Criteria:

* Pregnant or lactating woman.
* Life expectancy < 3 months.
* Serious, uncontrolled, concurrent infection(s) or illness(es)
* Any prior oxaliplatin treatment, with the exception of adjuvant therapy given > 12 months prior to the beginning of study therapy
* Prior unanticipated severe reaction to fluoropyrimidine therapy, known hypersensitivity to 5-fluorouracil, or known DPD deficiency
* Prior unanticipated severe reaction or hypersensitivity to platinum based compounds.
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer.
* Current, recent (within 4 weeks of first infusion on this study) or planned participation in an investigational drug study.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) within the last 6 months.
* History of clinically significant interstitial lung disease and/or pulmonary fibrosis.
* History of persistent neurosensory disorder including but not limited to peripheral neuropathy.
* Presence of central nervous system or brain mets.
* Major surgery, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 109/L, platelet count < 100 x 109/L)
  * Urine protein: creatinine ratio >/= 1.0 Impaired renal function with estimated creatinine clearance < 30 ml/min as calculated with Cockroft et Gault equation:
  * Serum bilirubin > 1.5 x upper normal limit. ALT, AST > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases)
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease)
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Blood pressure > 150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to Day 0.
* Serious, non-healing wound, ulcer or bone fracture
* Carcinoma of any histology in close proximity to a major vessel, cavitation or history of hemoptysis.
* Completion of previous adjuvant chemotherapy regimen < four weeks prior to the start of study treatment (within six weeks of study treatment for mitomycin C and nitroureas), or with related toxicities unresolved prior to the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-02; Primary Completion 2009-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C. Norris Comprehensive Cancer Center
Locations (1):
- U.S.C./Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Hurwitz H, Mitchell EP, Cartwright T, Kwok A, Hu S, McKenna E, Patt YZ. A randomized, phase II trial of standard triweekly compared with dose-dense biweekly capecitabine plus oxaliplatin plus bevacizumab as first-line treatment for metastatic colorectal cancer: XELOX-A-DVS (dense versus standard). Oncologist. 2012;17(7):937-46. doi: 10.1634/theoncologist.2012-0071. Epub 2012 May 23. PMID 22622147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this trial opened in February 2005 and closed in May 2009. All subjects were seen at USC.
Pre-assignment Details: This trial has no pre-assignment. All subjects were given the same treatment.
Groups:
- Oxaliplatin Followed by Bevacizumab, With Capecitabine: oxaliplatin 85 mg/m2 q 14 days, followed by bevacizumab 5 mg/kg q 14 days, with capecitabine 750 mg/m2 bid daily
Period: Overall Study
Arm/Group | Oxaliplatin Followed by Bevacizumab, With Capecitabine
Started | 63
Completed | 53
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lack of Efficacy | 8

BASELINE CHARACTERISTICS:
Population: All the participants who were enrolled are included in the analysis as per protocol.
Arm/Group | Oxaliplatin Followed by Bevacizumab, With Capecitabine
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Median Time for Progression Free Survival
Description: Progression-free survival was measured from the start of treatment until the time the subject is first recorded as having disease progression (progression = 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed or baseline, progression of non-measurable disease in the opinion of treating physician, appearance of new lesion/site, death due to disease), or death due to any cause. If a subject has not progressed or died, progression-free survival was censored at the time of last follow-up or the start of another treatment, whichever came first.
Time Frame: Up to 6 years
Population: All enrolled participants who receive the first course of treatment are included in the analysis as per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oxaliplatin Followed by Bevacizumab, With Capecitabine
Number analyzed (Participants) | 63
Months | 15.8 [11.5 to 64.3]

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Toxicity
Description: Summary of grade 3 (per CTCAE v3.0) or higher toxicities which generally is described as a severe adverse reaction or symptom.
Time Frame: Baseline, every 2 weeks of each cycle, and at end of treatment, up to 18 months.
Population: All enrolled participants who receive the first course of treatment are included in the analysis as per protocol.
Measure: Number; unit: Participants
Arm/Group | Oxaliplatin Followed by Bevacizumab, With Capecitabine
Number analyzed (Participants) | 63
Participants | 51

ADVERSE EVENTS:
Time Frame: Baseline, every 2 weeks of each cycle, and treatment end, up to 18 months.
Groups:
- Oxaliplatin Followed by Bevacizumab, With Capecitabine: oxaliplatin 85/m2 q 14 days, followed by bevacizumab 5 mg/kg q 14 days, with capecitabine 750 mg/m2 bid daily
Arm/Group | Oxaliplatin Followed by Bevacizumab, With Capecitabine
Serious Adverse Events (participants affected / at risk) | 51/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin Followed by Bevacizumab, With Capecitabine (N=63)
Alkaline phosphatase (Investigations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (7)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 3 (3)
Colitis, infectious (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Death not associated with CTCAE term (Death NOS) (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 17 (22)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (6)
Febrile neutropenia (fever, unknown origin w/o clinically or microbiologically documented infection) (Blood and lymphatic system disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (3)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage, GI (colon) (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Infection with unknown ANC (Wound) (Infections and infestations) | 1 (1)
Lipase (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Neuropathy: sensory (Nervous system disorders) | 13 (16)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (2)
Obstruction, GU (Ureter) (Renal and urinary disorders) | 1 (1)
Pain (Abdomen NOS) (Gastrointestinal disorders) | 8 (10)
Pain (Bone) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Rectum) (Gastrointestinal disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 13 (15)
Thrombosis/thrombus/embolism (Injury, poisoning and procedural complications) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin Followed by Bevacizumab, With Capecitabine (N=63)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 19 (30)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4 (4)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 20 (31)
Amylase (Investigations) | 1 (1)
Anorexia (Gastrointestinal disorders) | 34 (47)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 27 (53)
Bilirubin (hyperbilirubinemia) (Investigations) | 22 (35)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 33 (57)
Creatinine (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 37 (82)
Dizziness (Nervous system disorders) | 2 (2)
Edema: limb (General disorders) | 5 (5)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 52 (98)
Fever (in absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 25 (47)
Hail loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 55 (107)
Hemorrhage, GI (Anus) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI (Oral cavity) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI (Rectum) (Gastrointestinal disorders) | 4 (4)
Hemorrhage, GI (Upper GI NOS) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU (Urinary NOS) (Renal and urinary disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Nose) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypertension (Vascular disorders) | 19 (26)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (2)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration (Depression) (Psychiatric disorders) | 3 (3)
Mucositis/stomatitis (Oral cavity) (Gastrointestinal disorders) | 21 (28)
Nail changes (Skin and subcutaneous tissue disorders) | 26 (32)
Nausea (Gastrointestinal disorders) | 41 (73)
Neuropathy: sensory (Nervous system disorders) | 59 (147)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 18 (31)
Pain (Abdomen NOS) (Gastrointestinal disorders) | 42 (74)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Chest/thorax NOS) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Head/headache) (Nervous system disorders) | 9 (16)
Pain (Muscle) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Rectum) (Gastrointestinal disorders) | 2 (3)
Platelets (Investigations) | 21 (32)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 23 (31)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 50 (110)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 2 (2)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 18 (31)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes